CLINICAL TRIAL: NCT04163809
Title: The Role of Virtual Reality During Regional Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Mary Vijjeswarapu, Physician, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00055672
Record Dates: First submitted 2019-11-03; First posted 2019-11-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Pain
Keywords: virtual reality; anxiety; pain; regional anesthesia
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Group (no VR) (No Intervention): Patients will be randomly allocated to the control group, which receives no Virtual Reality (VR) during the regional anesthesia procedure.
- Experimental Group (VR) (Experimental): Patients will be randomly allocated to the the experimental group, which receives VR during the regional anesthesia procedure.
  Interventions: Device: Virtual Reality with Oculus Go headset

INTERVENTIONS:
Device: Virtual Reality with Oculus Go headset — The investigator will place the Oculus Go VR headset on the patient. VR will provide distracting, pleasant visual stimulus from the beginning of the procedure (while the patient is being cleaned and draped) and removed immediately after the regional anesthesia procedure is complete for roughly 10-20 minutes. All patients receiving VR will view the same scene.
  Other Names: Oculus Go
  Arms: Experimental Group (VR)

SUMMARY:
In this study, we will analyze the role of virtual reality in acute pain and anxiety management for regional anesthesia in pre-operative patients at Cedars-Sinai Medical Center.

DETAILED DESCRIPTION:
Virtual reality (VR) is a technology that allows people to be immersed in an artificial 3D environment with visual and auditory stimulation. Recently, VR technology has been integrated into medical practices and used during multi-modal pain management. The purpose of this study is to analyze the role of VR in acute pain and anxiety management for regional anesthesia in pre-operative patients at Cedars-Sinai Medical Center (CSMC). Little is known about the role of virtual reality during regional anesthesia. Patients who volunteer to be apart of this study will be randomly assigned to one of two groups: one that receives VR (experimental group) and one that does not receive VR (control group) during the regional anesthesia procedure. Those who wear the Oculus Go virtual reality headset will view pleasant, distracting scenes. Patients that are included in the study must be between 18-64 years of age, pre-operative at CSMC, receiving regional anesthesia, and able to provide informed consent. No further follow up is required. Traditionally, pre-operative patients at CSMC do not have the option of wearing the VR apparatus during nerve block procedures, and some patients may receive pre-medications before nerve blocks. Those enrolled in the study will not receive pre-medication. Before and after the procedure, the patients will receive a brief questionnaire that will be used to determine if virtual reality can be an efficacious tool in reducing pain and anxiety during regional anesthesia. All data collection and storage will be at CSMC. If VR is found to have a statistically significant reduction of acute pain compared to the control group, we can offer VR to patients to help alleviate acute pain, discomfort, and anxiety during regional anesthesia procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Elective pre-operative patients at Cedars-Sinai Medical Center who are receiving regional anesthesia
2. Between ages 18-64
3. Patient must be able to provide informed consent

Exclusion Criteria:

1. Patients under the age of 18 & above age 64
2. Visual impairment
3. Pregnant women
4. Diagnosis of epilepsy/seizures, dementia, and/or cognitive impairment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Anxiety Level Prior to Regional Anesthesia | questionnaire given within 1 hour prior to regional anesthesia procedure
  questionnaire to rate anxiety on a scale of 0-10
Anxiety Level During Regional Anesthesia | questionnaire given within 1 hour after regional anesthesia procedure
  questionnaire to rate anxiety on a scale of 0-10
Pain Level Prior to Regional Anesthesia | questionnaire given within 1 hour prior to regional anesthesia procedure
  questionnaire to rate pain on a scale of 0-10
Pain Level During Regional Anesthesia | questionnaire given within 1 hour after regional anesthesia procedure
  questionnaire to rate pain on a scale of 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Mary Vijjeswarapu, MD, Principal Investigator — CSMC Department of Anesthesiology
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Das DA, Grimmer KA, Sparnon AL, McRae SE, Thomas BH. The efficacy of playing a virtual reality game in modulating pain for children with acute burn injuries: a randomized controlled trial [ISRCTN87413556]. BMC Pediatr. 2005 Mar 3;5(1):1. doi: 10.1186/1471-2431-5-1. PMID 15745448
- [Background] McCaul KD, Malott JM. Distraction and coping with pain. Psychol Bull. 1984 May;95(3):516-33. No abstract available. PMID 6399756
- [Background] Sharar SR, Alamdari A, Hoffer C, Hoffman HG, Jensen MP, Patterson DR. Circumplex Model of Affect: A Measure of Pleasure and Arousal During Virtual Reality Distraction Analgesia. Games Health J. 2016 Jun;5(3):197-202. doi: 10.1089/g4h.2015.0046. Epub 2016 May 12. PMID 27171578
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307